CLINICAL TRIAL: NCT06490692
Title: Ffect of Blood Flow Restriction Training on Lateral Epicondylitis Parameters in Patients With Tennis Elbow
Brief Title: The Effect of Blood Flow Restriction Training on Tennis Elbow
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed ElMelhat, Associate Professor of Physical Therapy, Beirut Arab University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: BFR Training
Record Dates: First submitted 2024-06-29; First posted 2024-07-08 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-06

CONDITIONS: Tennis Elbow; Lateral Epicondylitis; Lateral Epicondylitis, Unspecified Elbow
Keywords: blood flow restriction training; lateral epicondylitis; tennis elbow
MeSH Terms: conditions — Tennis Elbow | interventions — Blood Flow Restriction Therapy

STUDY DESIGN:
Intervention Model Description: A randomized controlled clinical trial.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Blood Flow Restriction Training Group (Experimental): The experimental group will undergo conventional physical therapy including ultrasound, stretching, icing, heat, and deep friction massage applied at the extensor origin. In addition, the experimental group will undergo blood flow restriction strength training including the following: the weight of the dumbbell should be between 20-40% of their 1 rep max. The exercises were targeting the extensor muscles, applied by extending the wrist while holding the dumbbel and exercises targeting the supinator's and pronators while the participants were holding the dumbbell with forearm in neutral position, and were asked to supinate or pronate their forearm.
  The cuff will be placed proximally at the affected arm and inflated to achieve 40% limb occlusion depending on size attested using a a golden standard vascular dopler and all blood flow restriction activities were done with a licensed and experienced physical therapist.
  Interventions: Other: Blood Flow Restriction Training
- Conventional Strength Training Group (Active Comparator): The active comparator group will undergo the same interventions as the experimental group with the addition of conventional strength training including the same program as the experimental group but without blood flow restriction of any kind: the weight of the dumbbell should be between 20-40% of their 1 rep max. The exercises were targeting the extensor muscles, applied by extending the wrist while holding the dumbbell for 4 sets (35 repetitions, 15 repetitions,15 repetitions,15 repetitions) respectively, and exercises targeting the supinator's and pronators while the participants were holding the dumbbell with forearm in neutral position, and were asked to supinate or pronate their forearm.
  Interventions: Other: Conventional Strength Training

INTERVENTIONS:
Other: Blood Flow Restriction Training — The affected limb will have a cuff placed proximally and inflated to occlude the blood flow by 40% attested using a golden standard vascular doppler after which the individuals will perform the strengthening program set forth by the physical therapist. This is preceded by other tennis elbow interventions such as ultrasound, stretching, and deep friction massage at the extensor origin.
  Arms: Blood Flow Restriction Training Group
Other: Conventional Strength Training — The individuals in this group will undergo the same conventional physical therapy program as the other group including ultrasound, stretching, and deep friction massage. In addition, they will undergo the same strengthening program set forth by the physical therapist however with no blood flow restriction of any kind.
  Arms: Conventional Strength Training Group

SUMMARY:
The goal of this randomized controlled clinical trial is to investigate the effects of blood flow restriction training on the parameters surrounding tennis elbow afflicted patients including pain, disability, and grip strength.

The main question this study aims to answer is:

1- Does blood flow restriction training offer significantly better effects on pain, disability, and grip strength when compared to conventional strength training without blood flow restriction in patients afflicted with tennis elbow? Research will compare two groups with tennis elbow where both will perform the same rehabilitation program consisting of conventional physical therapy for tennis elbow as well as a strength training program with the only difference being that one group will undergo blood flow restriction training while the other will not.

DETAILED DESCRIPTION:
Lateral epicondylitis, commonly known as Tennis elbow, is a musculoskeletal condition characterized by pain at the lateral epicondyle due to repetitive forearm and hand movements. While it often improves over time, some cases may worsen. Diagnosis involves physical signs, including pain, decreased grip strength, tenderness, and pain during wrist flexion. Medical imaging such as MRI and clinical tests like Mills and Cozen's are used for confirmation.

According to Lenoir, Mares, Carlier (2019), physical therapy is the primary treatment, with exercises like eccentric muscle strengthening, deep friction massage, stretching, ultrasound, and laser therapy proving beneficial. Blood flow restriction training (BFR) has gained interest for enhancing strength and muscle mass. BFR involves partially restricting blood flow using a strap or cuff, inducing muscle hypoxia. Despite the unclear mechanism, BFR has shown positive effects on muscle tissue, possibly related to hypoxia and muscular acidosis.

The lack of studies on BFR's impact, especially on smaller muscle groups like fingers and wrists, creates a need for investigation. Given the commonality and impact of lateral epicondylitis symptoms, this study aims to compare the effectiveness between BFR training with standard PT exercises and standard PT alone in patients with lateral epicondylitis. Thus the purpose of this study is to prove that BFR training is more effective than standard physical training in improving the parameters surrounding tennis elbow.

The participants will be randomized into 2 groups. The standard physical therapy (group1) training consists of :1-ultrasound therapy, 2-laser, 3-deep friction massage followed by ice on the proximal attachment of the extensor tendon, 4-heat, 5-stretching of the wrist flexors and extensors, 6-strengthing of the wrist extensors combined with BFR.

(Group 2) will be treated with the same interventions excluding BFR training. Participants in both groups will be receiving treatment 2 times per week for 12 sessions.

ELIGIBILITY:
Inclusion Criteria:

* Patients that were included in this study were diagnosed with lateral epicondylitis by a medical doctor for less than 3 months.
* Dominant hand was diagnosed with lateral epicondylitis.
* They were aged between 20 and 40 years old.
* With decreased grip strength and wrist range of motion.
* No history of physical therapy treatment for lateral epicondylitis for at least 6 months.

Exclusion Criteria:

* Patients with chronic diabetes.
* Any type of trauma or fracture in the upper extremities in the last 3 months.
* Patients with any vestibular problems.
* Patients with deep vein thrombosis (DVT).
* Patients with hypertension.
* Patients with cancer.

Ages: 18 Years to 28 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-06-29 (Actual); Primary Completion 2024-10-25 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
Hand Grip Strength | Taken initially before intervention process and after the conclusion of the intervention period (6 weeks, 12 sessions).
  The hand grip strength was tested using a Camry Dynamometer, which is a smedly spring type dynamomter, whose reliability and validity in measuring handgrip strength has been reported by available literature.

SECONDARY OUTCOMES:
Patient Related Tennis Elbow Evaluation Scale (PRTEES) | Taken initially before intervention process and after the conclusion of the intervention period (6 weeks, 12 sessions).
  A scale specifically developed for Lateral Epicondylitis and it was used to determine forearm pain and disability, this scale consists of two parts, namely pain (5 items) and functional activities (10 items), each item has a score from 0 (no pain at all when performing a task) to 10 (the worst pain or unable to perform the task). The total score is the combined score of the 2 parts (OZMEN, KOPARAL, KARATAS... et al 2021), and it is proven that it is a reliable and valid tool for measuring pain and disability in LE patients (Jafarian, Barati, Sadeghi-Demneh 2021)
Numerical Pain Rating Scale (NPRS) | Taken initially before intervention process and after the conclusion of the intervention period (6 weeks, 12 sessions).
  A widely used 11-point scale (0-no pain, 10- sever pain) which has been proven to have good test reliability in individuals with chronic pain (Cheatham, Stull, Kobler 2018)

CONTACTS AND LOCATIONS:
Locations (1):
- Beirut Arab University, Beirut, Lebanon

IPD SHARING:
Plan to Share IPD: Undecided